CLINICAL TRIAL: NCT06781320
Title: Digital Occlusal Analysis and Enamel Wear Assessment in Temporomandibular Disorder Patients Treated with Fully Digital Versus Conventional Stabilization Splints: a Randomized Controlled Clinical Trial
Brief Title: Digital Occlusal Analysis and Enamel Wear Assessment in Temporomandibular Disorder Patients Treated with Fully Digital Versus Conventional Stabilization Splints
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Sawi Mohamed, Dr, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112/498
Record Dates: First submitted 2024-12-30; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: TMD; Temporomandibular Disorders (TMD)
Keywords: temporomandibular disorder, TMD,; Digital occlusal analysis; enamel wear assessment; stabilization splints
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fully Digital Stabilization Splint (FD-SS) (Experimental): Description:
  Participants in this group will receive a stabilization splint fabricated using a fully digital workflow. The intervention includes:
  * Intraoral scanning of the maxillary and mandibular arches to create a digital model.
  * Jaw tracking using the Zebris JMA system to record mandibular movements.
  * CAD design of the splint using Exocad software.
  * Fabrication: 3D printing technology to manufacture the splint.
  Purpose:
  The FD-SS is designed to provide optimal occlusal stabilization, reduce TMJ stress, and minimize enamel wear over a 6-month period.
  Device Name: Fully Digital Stabilization Splint (FD-SS)
  Interventions: Device: stabilization splint
- Conventional Stabilization Splint (C-SS) (Active Comparator): Description:
  Participants in this group will receive a stabilization splint fabricated using conventional methods. The intervention includes:
  * Taking alginate impressions of the maxillary and mandibular arches to create plaster casts.
  * Jaw registration using a Lucia jig and a semi-adjustable articulator for occlusal adjustment.
  * Manual fabrication of the splint using polymethyl methacrylate (PMMA) resin.
  Purpose:
  The C-SS is designed to achieve occlusal stabilization and provide symptom relief for patients with temporomandibular disorders (TMD) over 6 months.
  Device Name: Conventional Stabilization Splint (C-SS)
  Interventions: Device: stabilization splint

INTERVENTIONS:
Device: stabilization splint — the patients will receive a stabilization splint fabricated using a fully digital workflow includes:
  Intraoral scanning of maxillary and mandibular arches to create a digital model.
  Jaw tracking using the Zebris JMA system to record mandibular movements. CAD design of the splint using Exocad software. Fabrication of the splint via 3D printing technology. The FD-SS is designed to provide optimal occlusal stabilization, reduce TMJ stress, and minimize enamel wear over 6 months.
  Or the patient will receive stabilization splint fabricated using conventional methods. The intervention includes:
  Taking alginate impressions of maxillary and mandibular arches to create plaster casts.
  Jaw registration using a Lucia jig and semi-adjustable articulator for proper occlusal adjustment.
  Manual fabrication of the splint using polymethyl methacrylate (PMMA) resin. The C-SS is designed to achieve occlusal stabilization and symptom relief for TMD patients over 6 months.

SUMMARY:
This randomized controlled research aimed to analyse the occlusion and assist the enamel wear before and after using of the stabilization splints produced by the conventional methods with the fully digitally fabricated stabilization splints.

Research question: Will the fully digital stabilization splint offer significantly better occlusal equilibration and enamel wear compared to the conventional stabilization splint? the primary outcome will be Digital occlusal analysis, and secondary outcome will be enamel wear assessment

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the effectiveness of fully digitally fabricated stabilization splints (FD-SS) versus conventionally manufactured stabilization splints (C-SS) in patients with temporomandibular disorders (TMD). The study focuses on two primary outcomes: digital occlusal analysis and enamel wear assessment over a 6-month period.

Participants are TMD patients aged 18-40 with stable jaw relations and intact dentition, randomly assigned (1:1) to the FD-SS or C-SS group. Digital occlusal analysis is performed using OccluSense technology, which captures bite force distribution and contact points dynamically and statically. Enamel wear is assessed quantitatively using an intraoral scanner paired with Geomagic Control X 3D software for surface matching analysis. Baseline and follow-up STL datasets are compared to quantify volumetric enamel loss with micrometer precision.

In the FD-SS group, fully digital stabilization splints are fabricated using a digital workflow that includes intraoral scanning, jaw tracking with Zebris JMA devices, and CAD/CAM design in Exocad software. Splints are manufactured using 3D printing technology. In the C-SS group, conventional splints are fabricated using alginate impressions, plaster casts, and manual adjustments on a semi-adjustable articulator.

This study aims to advance the understanding of digital technologies in managing TMD, providing evidence for their efficacy in improving occlusal balance and minimizing enamel wear.

ELIGIBILITY:
Inclusion Criteria:

1. 18-40 years old
2. complete dentition
3. intact tooth
4. no occlusal disorder
5. stable jaw relation
6. No ongoing dental therapy, such as orthodontic or prosthodontics treatment.

Exclusion Criteria:

1. pregnant/lactating women
2. temporomandibular joint lesions found on clinical palpation or medical imaging examination
3. dentoalveolar pathology or ongoing treatment related to TMD
4. jaw opening less than 3 fingers
5. patients with occlusal dysfunctions
6. Patients with severe or moderate periodontitis.
7. Unable to undergo examination or treatment due to the presence of a psychological or mental disorder.
8. Severe jaw functional limitations.
9. Removable dentures or partially dentate patients
10. Trauma of recent date towards face, head or neck

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-26 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
1. Occlusal Force Measurement: • Measured using OccluSense in Newtons (N). | 6 months
  Occlusal Force Measurement:
  * Measured using OccluSense in Newtons (N)

SECONDARY OUTCOMES:
Tooth Wear Measurement using an intraoral scanner | 6 months
  Comparison of STL datasets using Geomagic Control X software.
  * Measured as % of surface overlap or deviation in microns.

IPD SHARING:
Plan to Share IPD: Yes